CLINICAL TRIAL: NCT00725348
Title: An Open-Label, Multi-Center Pilot Trial to Assess the Efficacy and Safety of Oral R115866 in the Treatment of Subjects With Moderate to Severe Plaque Type Psoriasis
Brief Title: An Open-Label, Multi-Center Trial in the Treatment of Subjects With Moderate to Severe Plaque Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT0700NED001
Record Dates: First submitted 2008-07-17; First posted 2008-07-30 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2008-07

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — R 115866

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): R115866
  Interventions: Drug: Talarozole

INTERVENTIONS:
Drug: Talarozole — 1.0 mg oral dose per day
  Other Names: Rambazole; R115866

SUMMARY:
This is a study of a new oral drug used for the treatment of psoriasis. All subjects will get active medication, there is no placebo arm.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential (at least 2 years post-menopausal or undergone successful surgical sterilization at least 1 year before inclusion)
* Presence of moderate to severe plaque psoriasis with a PASI of at least 5

Exclusion Criteria:

* Pustular, guttate or other non-plaque forms of psoriasis or psoriatic arthritis
* Significant coexisting hepatic, renal, or bone marrow disease, hyperlipidemia, chronic pancreatitis, osteoporosis, or a history indicating adrenal cortex dysfunction or any other serious disease (including cancer and subjects known to be HIV positive)
* History of heart failure, myocardial infarction within the past six months, cardiac arrhythmia, or under treatment for heart disorders
* Clinically significant abnormal ECG-intervals or morphology of the ECG; QT or QTc >470 ms in females or >450 ms in males
* Use of vitamin A (>1000 µg/day), phenytoin, carbamazepine, warfarin, rifampicin, tetracyclines, ketoconazole, itraconazole, astemizole, terfenadine, cisapride, anti-psychotics, anti-depressants, lithium, antimalarials, alpha-blocking drugs, angiotensin-converting enzyme inhibitors, cyclosporin A, glucocorticosteroids and non-steroidal anti-inflammatory drugs, non-potassium-sparing diuretics
* Previous use of any systemic immunomodulatory therapy (biologicals) or psoriasis vaccine
* Use of other systemic therapy for psoriasis (e.g. PUVA, systemic steroids, cyclosporin A, methotrexate, retinoids) within four weeks prior to Visit 2
* Use of UV therapy or excessive UV exposure or topical therapy for psoriasis other than bland emollients within two weeks prior to Visit 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-04; Primary Completion 2005-03 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
PASI Scores | Various Visits

CONTACTS AND LOCATIONS:
Overall Officials: Prof. P. van de Kerkhof, MD, PhD, Principal Investigator — University of Nijmegen, Maastricht, The Netherlands
Locations (2):
- Netherlands (2):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum Nijmegen Sint Radboud, Nijmegen